CLINICAL TRIAL: NCT00646087
Title: Ketamine Frequency Treatment for Major Depressive Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Pilot study determined that this study would not be feasible.
Sponsor: Essentia Health (Other)
Responsible Party: Micheal Messer MD, St. Mary's Duluth Clinic Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-07-04
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (6K) (Experimental): 6K: 6 ketamine injections (0.5 mg/kg of ketamine) every other day for 12 days
  Interventions: Drug: Ketamine
- Ketamine/Placebo (2K4P) (Active Comparator): 2K4P = two active ketamine injections(2K) and four placebo (saline) injections over 12 days.
  Interventions: Drug: Ketamine/Saline

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg of ketamine every other day for 12 days (days 1, 3, 5, 7, 9, 11)
  Arms: Ketamine (6K)
Drug: Ketamine/Saline — 0.5 mg/kg of ketamine on days 1 and 7, placebo (saline) on days 3, 5, 9, 11
  Arms: Ketamine/Placebo (2K4P)

SUMMARY:
Depression is a wide spread illness. Depression contributes most significantly to national health care costs. While the number and types of treatments used for depression have expanded over the years, even with an increased range of options, the response rate, defined as the number of subjects who have a 50% reduction in depressive symptoms, is estimated to be around 65%.

This randomized clinical trial will examine the frequency of treatment with ketamine in patients with treatment-resistant depression TRD without psychosis. It will compare two modes of the ketamine treatment; every other day ketamine, versus two active and four placebo treatments over the period of 12 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65
* Major depressive disorder without psychotic features confirmed by a structured clinical diagnostic interview, SCID.
* Treatment resistant depression defined using the Antidepressant Treatment History Form (ATHF)
* HDRS 21 score > 18
* Female participants of childbearing potential must be using a medically accepted means of contraception (birth control pills, spermicidal barrier)
* Ability to concur with medication standardization regiment (section as an outpatient
* Physically healthy (no chronic diseases; normal CBC, BMP, AST, ALT, and UA)
* Competent to give informed consent to all required tests and examinations and sign a consent document

Exclusion Criteria:

* Bipolar disorder
* Psychosis or any other psychotic disorder as defined by DSM-IV criteria
* Serious or imminent threat for suicide
* Pregnant or nursing female
* Presence of serious unstable medical illnesses including hepatic, renal, gastrointestinal, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, or abnormal laboratory tests (CBC, BMP, AST, ALT, and UA)
* Uncontrolled hypertension
* History of CVA
* Treatment with St. Johns wort, tramadol, phentolamine, naloxone, or anticholinergic medications
* Alcohol or illicit drug abuse for 6 months (evidence from UDS)
* Currently involved in a clinical trial or used an experimental medication within the last 30 days
* Hypersensitivity to ketamine products

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03

PRIMARY OUTCOMES:
The primary efficacy measure is the change in scores in the 21-item Hamilton Depression Rating Scale. | 20 weeks

SECONDARY OUTCOMES:
Proportion of patients with remission (HDRS score < 18) at the end of the 2-week treatment and each follow-up contact. | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Messer, MD, Principal Investigator — Essentia Health
Locations (1):
- St. Mary's Duluth Clinic Health System, Duluth, Minnesota, United States

REFERENCES:
- [Background] Pincus HA, Pettit AR. The societal costs of chronic major depression. J Clin Psychiatry. 2001;62 Suppl 6:5-9. PMID 11310818
- [Background] Holtzheimer PE 3rd, Nemeroff CB. Advances in the treatment of depression. NeuroRx. 2006 Jan;3(1):42-56. doi: 10.1016/j.nurx.2005.12.007. PMID 16490412
- [Background] Nierenberg AA, Amsterdam JD. Treatment-resistant depression: definition and treatment approaches. J Clin Psychiatry. 1990 Jun;51 Suppl:39-47; discussion 48-50. PMID 2112132
- [Background] Burrows GD, Norman TR, Judd FK. Definition and differential diagnosis of treatment-resistant depression. Int Clin Psychopharmacol. 1994 Jun;9 Suppl 2:5-10. doi: 10.1097/00004850-199406002-00002. PMID 7930496
- [Background] Crown WH, Finkelstein S, Berndt ER, Ling D, Poret AW, Rush AJ, Russell JM. The impact of treatment-resistant depression on health care utilization and costs. J Clin Psychiatry. 2002 Nov;63(11):963-71. doi: 10.4088/jcp.v63n1102. PMID 12444808
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Correll GE, Futter GE. Two case studies of patients with major depressive disorder given low-dose (subanesthetic) ketamine infusions. Pain Med. 2006 Jan-Feb;7(1):92-5. doi: 10.1111/j.1526-4637.2006.00101.x. No abstract available. PMID 16533209
- [Background] Kudoh A, Takahira Y, Katagai H, Takazawa T. Small-dose ketamine improves the postoperative state of depressed patients. Anesth Analg. 2002 Jul;95(1):114-8, table of contents. doi: 10.1097/00000539-200207000-00020. PMID 12088953
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Hirota K, Lambert DG. Ketamine: its mechanism(s) of action and unusual clinical uses. Br J Anaesth. 1996 Oct;77(4):441-4. doi: 10.1093/bja/77.4.441. No abstract available. PMID 8942324
- [Background] Paul IA, Skolnick P. Glutamate and depression: clinical and preclinical studies. Ann N Y Acad Sci. 2003 Nov;1003:250-72. doi: 10.1196/annals.1300.016. PMID 14684451
- [Background] Annetta MG, Iemma D, Garisto C, Tafani C, Proietti R. Ketamine: new indications for an old drug. Curr Drug Targets. 2005 Nov;6(7):789-94. doi: 10.2174/138945005774574533. PMID 16305457
- [Background] Stewart CE. Ketamine as a street drug. Emerg Med Serv. 2001 Nov;30(11):30, 32, 34 passim. PMID 11759641
- [Background] Correll GE, Maleki J, Gracely EJ, Muir JJ, Harbut RE. Subanesthetic ketamine infusion therapy: a retrospective analysis of a novel therapeutic approach to complex regional pain syndrome. Pain Med. 2004 Sep;5(3):263-75. doi: 10.1111/j.1526-4637.2004.04043.x. PMID 15367304
- [Background] Leonard B. Clinical implications of mechaniszms of action of antidepresants. Advan Psychiatr Treat. 2000;6:178-186.
- [Background] Beck AT, Beamesderfer A. Assessment of depression: the depression inventory. Mod Probl Pharmacopsychiatry. 1974;7(0):151-69. doi: 10.1159/000395074. No abstract available. PMID 4412100
- [Background] Beck AT, Steer RA, Garbin MG. Psycometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clin Psychol Rev. 1988;8:77-100.
- [Background] Overall J, Gorham D. The brief psychiatric rating scale. Psycol Rep. 1962;10:799-812.
- [Background] Bremner JD, Krystal JH, Putnam FW, Southwick SM, Marmar C, Charney DS, Mazure CM. Measurement of dissociative states with the Clinician-Administered Dissociative States Scale (CADSS). J Trauma Stress. 1998 Jan;11(1):125-36. doi: 10.1023/A:1024465317902. PMID 9479681
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] First MB, Spitzer RL, Miriam G, Williams JBW. Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Patient Edition. (SCID-I/P). New York: Biometrics Research, New York State Psychiatric Institute; 2002